CLINICAL TRIAL: NCT04609358
Title: Efficacy and Safety of the Implementation of an Algorithm for Enteral Nutrition Support Compared With Traditional Practice in Children With Congenital Heart Disease: Randomized Clinical Trial, Simple Blind.
Brief Title: Efficacy and Safety of the Algorithm for Enteral Nutrition Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xu Zhuoming, Director of CICU, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: SCMCIRB-K2015003
Record Dates: First submitted 2017-04-04; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Nutrition Disorder, Child
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The patients' nutrition were supported according the the algorithm of the enteral nutrition.
  Interventions: Other: intervention group
- Control group (No Intervention): The patients' nutrition were supported according the prescription of the physicians and dietician in our hospital.

INTERVENTIONS:
Other: intervention group — When patients' hemodynamics was stable, start 1-2ml/kg/hr post-op 6-12 hours and increased 1-2ml/kg/hr each day if tolerating to reach the target energy supply When patients' hemodynamics wasn't stable, start post-op 6-12 hours 0.5-1ml/kg/hr and increased 0.5-1ml/kg/hr each day if tolerating to reach the target energy supply.
  Arms: Intervention group

SUMMARY:
The purpose of this trial is to evaluate the efficacy and safety of the implementation of an algorithm for enteral nutrition support compared with usual standard practice in children with malnutrition status with congenital heart disease

DETAILED DESCRIPTION:
In many developing countries, pediatric cardiac programs are not fully established, and nutrition support algorithm is lack. Therefore, this study aimed to evaluate the the efficacy and safety of the implementation of an algorithm for enteral nutrition support compared with usual standard practice in children with malnutrition status with congenital heart disease. The usual standard practice for feeding often interrupted by retention in the gut and then choose the parenteral nutrition support especially in the patients with unstable hemodynamic status. Actually tiny and continuous feeding would improve the gut function and reach the adequate energy supply.

ELIGIBILITY:
Inclusion Criteria:

weight-for-age of z-score <-2; or length-for-age of z score <-2; or weight-for-length of z score <-2

Exclusion Criteria:

Any patient with congenital genetic metabolic diseases

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Malnutrition recovery | 1 year
  Malnutrition was assessed as recovering from malnutrition

SECONDARY OUTCOMES:
Feeding intolerance | 1 year
  According to the criteria established by the American Academy of Pediatrics in 2003, the following symptoms are diagnosed as feeding intolerance: severe abdominal distension or discoloration; Signs of intestinal perforation; Obvious blood stool; Gastric retention ≥ 25% of the total amount after 2 to 3 feeding intervals; Bile reflux or vomiting; Severe apnea or bradycardia; Severe cardiopulmonary insufficiency; Apnea: Cessation of breathing for ≥20 seconds, or cessation of breathing accompanied by a decrease in SpO2.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuoming Xu, PhD, Study Director — Shanghai Children's Medical Center
Locations (1):
- Cardiac intensive care unit, Department of cardiothoracic vascular surgery, Shanghai Children's Medical Center, Medical college of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Zhang M, Song Y, Luo Y, Wang L, Xu Z, Bao N. Early high-energy feeding in infants following cardiac surgery: a randomized controlled trial. Transl Pediatr. 2021 Oct;10(10):2439-2448. doi: 10.21037/tp-21-360. PMID 34765467